CLINICAL TRIAL: NCT04466995
Title: Factors Affecting Endotracheal Cuff Pressure in Laparoscopic and Laparotomic Gynecological Cases and Its Effect on Postoperative Respiratory Complications
Brief Title: Factors Affecting Endotracheal Cuff Pressure in Gynecological Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Güneş Özlem Yıldız, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020/92
Record Dates: First submitted 2020-06-05; First posted 2020-07-10 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Intubation Complication

STUDY DESIGN:
Intervention Model Description: Endotracheal tube pressure will be measured in the surgical technique using 2 different methods.(laparoscopic and laprotomic)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laparoscopic gynecologic surgery (Experimental): 25 laparoscopic surgery to endotracheal cuff pressure 5., 15., 30., 45. min will be measured, values will be recorded
  Interventions: Device: manometer
- laparotomic gynecologic surgery (Other): 25 laparotomic surgery to endotracheal cuff pressure 5., 15., 30., 45. min will be measured, values will be recorded
  Interventions: Device: manometer

INTERVENTIONS:
Device: manometer — cuff pressure to be measured with manometer

SUMMARY:
Postoperative airway complications associated with endotracheal intubation can be seen.

While some of these complications are predictable, some may occur urgently. If the endotracheal cuff is over-inflated and its pressure is high, mucosal damage resulting from mucosal pressure is one of the main factors for tracheal morbidity. Endotracheal tube cuff pressure is not routinely measured. It was confirmed that the palpation of the pilot balloon was insufficient to detect high cuff pressures. In laparoscopic cases, the investigators aimed to investigate whether the increase in intra-abdominal pressure as a result of carbon dioxide insufflation, and the change of respiratory functions after trendelenburg position are effective on cuff pressure and whether there is a difference compared to laparotomic cases.

DETAILED DESCRIPTION:
It was planned to include 50 patients in the American Anesthesiologists Association (ASA) 1-3 risk score group, which will be an elective gynecological operation between the ages of 18-70. When patients arrive in the operating room, after the ECG, pulse oximeter, non-invasive pressure monitoring is provided in the supine position, 18 gauge intravenous(iv) vascular access will be opened and balanced fluid 4-6 ml / kg / h will be inserted. Anesthesia induction with midazolam 0.05 mg / kg, propofol 2-3 mg / kg, Fentanyl 1-2 µg / kg and rocuronium 0.6 mg / kg will be achieved after 3 minutes of preoxygenation. he muscle relaxant effect will be monitored by monitoring TOF (train of four), and after sufficient relaxation (TOF 95%), the anesthetist will be intubated with the 7-7.5 number endotracheal tube suitable for the high-volume low-pressure patient. The cuff of the endotracheal tube will be inflated with the help of an injector and the cuff will be attached to the manometer. Cuff pressures will be inflated to 25 mmHg. The patients will be given oxygen at 40% and air at 3lt / min. The maintenance of anesthesia will be achieved with sevoflurane and 0.05-0.1mcg / kg / min remifentanil infusion.

If the patient feels pain in the perioperative period, 50 mcg fentanyl iv will be used as rescue analgesia. During the operation, rokurunium (0.2mg / kg) boluses will be delivered according to the patient's clinic and the TOF value between 0-2 (depending on the type of surgery). Mechanical ventilation will be started in volume controlled mode with 6-8 ml / kg tidal volume, and 12 frequencies. Respiratory frequencies,tidal volume and positive end expiratory pressure (PEEP) values of patients will be optimized so that end tidal CO2 is 35-45 mmHg throughout the case. At the end of surgery, 100 mg tramadol and 1 g paracetamol will be administered to patients for the purpose of postoperative analgesia. Patients will be extubated after the muscle relaxant is recurrentized with 0.03mg / kg neostigmine and 0.01mg / kg atropine.

If the patient's numeric rating scale (NRS) score is 3 or more during recovery, 0.3 mg / kg Petidine hydrochloride will be applied as rescue analgesia. The 'Case Tracking Form' prepared for the follow-up of the research will be recorded demographically, age, height, weight and BMI information of the patients in the preoperative period.

In the perioperative period, cuff pressures in the supine position after intubation, at the 5th, 15th, 30th, 45th minutes and before extubation will be measured and recorded with the cuff manometer. In addition to the follow-up form, intra-abdominal pressure, PEEP, P peak and P plateau values, anesthesia time, operation time during each measurement will be recorded. Patients who were followed-up in the recovery were evaluated by the service nurse who did not know how to work in the service at the postoperative 1st, 12th, 24th hours, and the NRS (numeric rating scale) (0 is painless, 10 is the most painful and will be asked to describe the pain from 1 to 10); It will be evaluated in terms of dysphagia, cough, sore throat, hoarseness.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18-70 years old who will undergo gynecological abdominal surgery
* Patients with American Society of Anesthesiologists physical status 1-3
* Patients who will undergo elective surgery

Exclusion Criteria:

* Patients with tracheotomy
* Patients with detected tracheal stenosis
* Patients with laryngeal disease or laryngeal surgery
* Patients with difficult airway (intubated after 2 or more attempts)
* Patients with BMI> 35
* Patients receiving chronic obstructive pulmonary disease treatment
* Patients with ASA ≥4

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
cuff pressure | 1 hour
  cuff pressure to be measured with manometer

CONTACTS AND LOCATIONS:
Overall Officials: gunes o yildiz, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)